CLINICAL TRIAL: NCT06643208
Title: Department of Hepatobiliary Pancreatic Surgery, Fujian Provincial Hospital
Brief Title: D-TACE-HAIC Combined With Envafolimab and Lenvatinib for Unresectable ICC
Status: Recruiting | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Mao-Lin Yan, Principal Investigator, Fujian Provincial Hospital
Other Study IDs: TALENP005
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — envafolimab; lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combination therapy group: Patients with unresectable cholangiocarcinoma were treated with D-TACE-HAIC (GEMOX regimen) combined with envafolimab and lenvatinib
  Interventions: Drug: TACE-HAIC, Envafolimab and Lenvatinib

INTERVENTIONS:
Drug: TACE-HAIC, Envafolimab and Lenvatinib — TACE-HAIC (GEMOX regimen) combined with Envafolimab and Lenvatinib

SUMMARY:
This is a prospective, single-arm, multicenter, phase II trial to evaluate the efficacy and safety of D-TACE-HAIC (GEMOX protocol) in combination with Envafolimab and Lenvatinib for unresectable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ages of 18 and 75;
* 2. Child-Pugh liver function grade: A/B;
* 3. ECOG score (see annex for scoring standards) : ≤1 score;
* 4. ICC was confirmed by pathology and evaluated by two senior hepatobiliary surgeons as unresectable for surgery (including multiple intrahepatic lesions, local vascular invasion, local lymph node metastasis, and distant metastasis);
* 5. According to RECIST 1.1 criteria, the patient has at least one measurable lesion (the CT/MRI scan diameter of the lesion can be measured ≥10mm, and the lesion has not received local treatment such as radiotherapy or freezing);
* 6. The expected survival time is greater than 3 months;
* 7. Patients who had not received any tumor-related targeting, immunization, radiotherapy or chemotherapy before enrollment;
* 8. Functional indexes of vital organs met the following requirements: · Routine blood: absolute neutrophil count ≥1.5×109/L, Hb≥9.0g/L, PLT≥75×109/L; · Liver function: total bilirubin ≤1.5 times the upper limit of normal (ULN) (≤2.5 times ULN after biliary drainage in patients with obstructive jaundice); Alanine aminotransferase (ALT), aspartate aminotransferase (AST)≤ 5x ULN, albumin ≥30g /L; · Renal function: serum creatinine ≤1.5mg/dL, creatinine clearance ≥60ml /min; · Coagulation function: International standardized ratio (INR) and activated partial thromboplastin time (APTT)≤1.5 times ULN;
* 9. No history of severe arrhythmia or heart failure; No history of severe ventilation dysfunction or severe pulmonary infection;
* 10. Women of childbearing age should agree to use contraception during the use of medication and for 6 months after the end of medication; Patients who had a negative serum or urine pregnancy test in the 7 days prior to study enrollment and must be non-lactating patients, men should consent to use contraception during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* 1. Patients who have previously received other local anti-tumor treatments (such as radiotherapy, radiofrequency ablation, etc.), who are allowed to relapse 6 months after previous surgery, and who are allowed to undergo biliary drainage (including PTCD and biliary stent implantation);
* 2. History of allergy to gemcitabine, oxaliplatin, Envolizumab, Renvastinib and its components;
* 3. A history of other malignant tumors within the past 5 years or at the same time, except cured basal cell carcinoma of the skin, cervical carcinoma in situ and thyroid papillary carcinoma;
* 4. Patients who have previously received an organ transplant or are planning to receive an organ transplant;
* 5. The presence of any active autoimmune disease or patients with autoimmune disease and expected recurrence (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes);
* 6. History of immune deficiency; The patient is taking immunosuppressants or systemic hormone therapy for immunosuppressive purposes and continues to use it within 2 weeks prior to signing the informed consent;
* 7. Known hereditary or acquired bleeding (e.g. coagulation disorders) or thrombotic tendencies, e.g. in hemophiliacs; Is currently or recently (within 10 days prior to the start of study therapy) used full dose oral or injectable anticoagulants or thrombolytic agents for therapeutic purposes (prophylactic use of low-dose aspirin, low-molecular weight heparin permitted);
* 8. Serious infections, such as severe pneumonia, bacteremia, and comorbiditis requiring hospitalization, occurred within 4 weeks prior to the first use of the study drug; Baseline chest imaging findings indicate active lung inflammation, signs and symptoms of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment (excluding prophylactic antibiotic use);
* 9. Patients with mental illness; Have a history of psychotropic substance abuse, alcoholism and drug use;
* 10. Pregnant or lactating women;
* 11. Those who, according to the judgment of the researcher, should not participate in this experiment for other reasons;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with unresectable intrahepatic cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | Four weeks after the initiation of medication
  The Objective response rate (ORR) was defined as the complete response (CR) rate or the partial response (PR) rate according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival, OS | From date of enrollment until the date of death from any cause, assessed up to 60 months
  The Overall survival (OS) was defined as the time between receiving treatment and observing death or loss of follow-up for any reason.
Progression-free survival, PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The Progression free survival (PFS) was defined as the time between the start of treatment and the progression of intrahepatic and/or extrahepatic tumors, or the occurrence of death or loss of follow-up for any reason.
Disease control rate, DCR | Four weeks after the initiation of medication
  The Disease control rate (DCR) was defined as the complete response (CR) rate or the partial response (PR) rate or stable disease (SD) rate according to RECIST v1.1 criteria.
Treatment-related adverse events, TRAEs treatment-related adverse events | From the initiation of medication, with recordings made whenever an adverse reaction occurs, assessed up to 12 months
  The incidence, spectrum and severity of adverse events (AE) and serious adverse events (SAE) were determined according to the NCI-CTCAE V5.0 standard. Dose suspension rate and dose termination rate due to adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Maolin Yan, Doctor, Study Chair — Department of Hepatobiliary Pancreatic Surgery, Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No